CLINICAL TRIAL: NCT01969123
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-Group, 26-Week, Phase 3 Study of 2 Doses of EVP-6124 or Placebo in Subjects With Mild to Moderate Alzheimer's Disease Currently or Previously Receiving an Acetylcholinesterase Inhibitor Medication
Brief Title: Study of the Safety and Effectiveness of Two Doses of Investigational Study Drug EVP-6124 in Subjects With Alzheimer's Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study has been suspended due to clinical hold.
Sponsor: FORUM Pharmaceuticals Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EVP-6124-024; 2013-002618-10 (EudraCT Number)
Record Dates: First submitted 2013-10-21; First posted 2013-10-25 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2015-09

CONDITIONS: Alzheimer's Disease; Dementia
Keywords: Alzheimer's disease; Cognition; Alpha-7 nAChR
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — 7-chloro-N-quinuclidin-3-yl-benzo(b)thiophene-2-carboxamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Experimental: EVP-6124, low dose (Experimental): low dose, Tablet, Once Daily, Day 1 through Day 182
  Interventions: Drug: Drug: EVP-6124
- Experimental: EVP-6124, high dose (Experimental): high dose, Tablet, Once Daily, Day 1 through Day 182
  Interventions: Drug: Drug: EVP-6124
- EVP-6124 Placebo (Placebo Comparator): Placebo, Tablet, Once Daily, Day 1 through Day 182
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Drug: EVP-6124
  Arms: Experimental: EVP-6124, high dose; Experimental: EVP-6124, low dose
Drug: Placebo
  Arms: EVP-6124 Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of 2 fixed doses of EVP-6124 compared to placebo for 26 weeks in subjects with mild to moderate Alzheimer's disease currently receiving stable treatment or previously treated with an acetylcholinesterase inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* Ages ≥55 and ≤85 years
* Informed consent form (ICF) signed by the subject or legally acceptable representative before any study-specific procedures for the subject are performed and an ICF signed by the support person/caregiver before any study-specific procedures for the support person/caregiver are performed
* Clinical diagnosis of dementia due to probable AD consistent with criteria established by a workgroup of the National Institute on Aging and the Alzheimer's Disease Association
* Clinical decline within 12 months before screening and onset of symptoms at least 12 months or longer before screening, which may include any documented cognition, functional, or other objective assessment or the clinical judgment of the investigator or the subject's referring physician that the subject has experienced a clinical decline within the last 12 months
* Magnetic resonance imaging (MRI) or computed tomography (CT) scan performed within 12 months before screening, with findings consistent with the diagnosis of dementia due to AD without any other clinically significant comorbid pathologies. If an MRI or CT scan is unavailable or occurred greater than 12 months before screening, this assessment should be completed and the findings confirmed before the subject enters the run-in period (Day -14) (copy of the report will be available at the study site)
* Mini-Mental State Examination (MMSE) score ≥14 and ≤24 at screening and confirmed on Day 1 prior to randomization (fluctuations of ±2 points are acceptable on Day 1/baseline)
* Clinical Dementia Rating Global score (CDR-GS) ≥1 (at least mild dementia) at screening and confirmed on Day 1 prior to randomization
* Modified Hachinski Ischemic Scale (mHIS) score ≤4 at screening
* Fertile, sexually active subjects (men and women) must use an effective method of contraception during the study. Female subjects and the female partner of male subjects must be surgically sterile (hysterectomy or bilateral tubal ligation), postmenopausal for at least 1-year, or willing to practice adequate methods of contraception if of childbearing potential (defined as consistent use of combined effective methods of contraception [including at least 1 barrier method])
* Reliable and capable support person/caregiver, who if not living in the same household, interacts with the subject approximately 4 times per week and will be available to attend clinic visits in person when possible
* Subject living at home, senior residential setting, or an institutional setting without the need for continuous (ie, 24-hour) nursing care
* General health status acceptable for participation in a 26-week study
* Fluency (oral and written) in the language in which the standardized tests will be administered
* Receiving a stable dose of an acetylcholinesterase inhibitor (AChEI) (donepezil, rivastigmine or galantamine) for at least 3 months (90 days) before screening and with continuous dosing for at least 6 months OR not presently receiving an AChEI (at least 30 days before screening), but with a history of previous AChEI treatment (subjects receiving donepezil 23 mg currently or within 3 months before screening are ineligible)

Exclusion Criteria:

* Exposure to an experimental drug, experimental biologic or experimental medical device within 2 months (60 days) before screening
* Prior participation in an amyloid vaccination clinical study at any time in the past or completion of a passive amyloid vaccination study within 6 months before screening
* Inability to swallow a tablet
* In the judgment of the investigator, inability of the subject or the support person/caregiver to complete a 26-week study
* Inability to be ≥75% compliant with single-blind study drug
* Inability to adequately cooperate or complete the cognitive testing procedures or any study assessment
* Residence in a skilled nursing facility
* Untreated vitamin B12 or folate deficiency (if treated, must be stably treated for at least 6 months before screening)
* Clinically significant (in the judgment of the investigator) abnormal serum electrolytes (sodium, potassium, magnesium) after repeat testing
* Clinically significant untreated hypothyroidism (if treated, thyroid-stimulating hormone level and thyroid supplementation dose must be stable for at least 6 months before screening)
* Insufficiently controlled diabetes mellitus (in the judgment of the investigator) or requiring insulin
* Renal insufficiency (serum creatinine >2.0 mg/dL)
* Malignant tumor within 3 years before screening (except squamous and basal cell carcinoma or cervical carcinoma in situ or localized prostate cancer)
* Female subjects who are pregnant, nursing, or planning to become pregnant during the study
* Unstable medical condition that is clinically significant in the judgment of the investigator
* Alanine transaminase (ALT) or aspartate transaminase (AST) >2.5 times the upper limit of normal
* History of myocardial infarction or unstable angina within 6 months before screening
* History of more than 1 myocardial infarction within 5 years before screening
* Clinically significant (in the judgment of the investigator) cardiac arrhythmia (including atrial fibrillation), cardiomyopathy, or cardiac conduction defect (subjects with a pacemaker are acceptable)
* Symptomatic hypotension or hypertension (supine diastolic blood pressure >95 mmHg) (in the judgment of the investigator)
* Clinically significant abnormality on screening or baseline electrocardiogram (ECG), including but not necessarily limited to a confirmed corrected QT interval (QTc) value ≥450 msec for males or ≥470 msec for females. In subjects with a QRS value >120msec, those with a QTc value <500 msec may be eligible following discussion with the Medical Monitor.
* Stroke within 18 months before screening, or history of a stroke concomitant with onset of dementia
* History of brain tumor, subdural hematoma, or other clinically significant (in the judgment of the investigator) space-occupying lesion on CT or MRI
* Head trauma with clinically significant (in the judgment of the investigator) loss of consciousness within 12 months before screening or concurrent with the onset of dementia
* Onset of dementia secondary (in the judgment of the investigator) to cardiac arrest, surgery with general anesthesia, or resuscitation
* Specific degenerative central nervous system (CNS) disease diagnosis other than AD (eg, Huntington's disease, Creutzfeld-Jacob disease, Down's syndrome, Fronto-Temporal Dementia, Parkinson's disease)
* Subjects with no history of prior treatment with an AChEI (donepezil, rivastigmine, or galantamine)
* Memantine currently or within 30 days before screening
* Antipsychotics; low doses (in the judgment of the investigator, except clozapine) are allowed only if given for sleep disturbances, agitation and/or aggression, and only if the subject has received a stable dose for at least 3 months before screening (but not within 8 hours before any cognitive test)
* Tricyclic antidepressants and monoamine oxidase inhibitors; all other antidepressants are allowed only if the subject has received a stable dose for at least 3 months before screening
* Antiepileptic medications if taken for control of seizures
* Chronic intake of opioid-containing analgesics
* Sedating H1 antihistamines
* Nicotine therapy (including the patch), varenicline (Chantix), or similar therapeutic agent within 30 days before screening
* Clinically significant urine drug screen or serum alcohol test result in the judgment of the investigator
* History of ischemic colitis or ischemic enterocolitis

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 474 (Actual)
Dates: Start 2013-10; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Alzheimer's Disease Assessment Scale-Cognitive Subscale 13-item (ADAS-Cog-13) to Day 182 | Baseline to Day 182 or Early Termination
Change from Baseline in the Clinical Dementia Rating Sum of the Boxes (CDR-SB) to Day 182 | Baseline to Day 182 or Early Termination
Safety and tolerability of EVP-6124 or Placebo in Subjects with AD | Baseline to Day 182 or ET
  All adverse experiences spontaneously reported by subject and/or observed by an investigator and repeated clinical evaluation of physical exam, vital signs, 12-lead ECG (electrocardiogram), ambulatory ECG and laboratory tests (hematology/blood chemistry/urinalysis)

SECONDARY OUTCOMES:
Change from Baseline in activities of daily living using the Disability Assessment for Dementia (DAD) | Baseline to Day 182 or Early Termination
Change from Baseline in psychiatric and behavioral symptoms using the Neuropsychiatric Inventory (NPI) | Baseline to Day 182 or Early Termination
Change from Baseline in the Mini-Mental State Examination (MMSE) | Baseline to Day 182 or Early Termination
Change from Baseline in the Controlled Oral Word Association Test (COWAT) | Baseline to Day 182 or Early Termination

CONTACTS AND LOCATIONS:
Locations (82):
- United States (44):
  - Phoenix, Arizona
  - Tucson, Arizona
  - Costa Mesa, California
  - Encino, California
  - Glendale, California
  - Long Beach, California
  - Redding, California
  - San Diego, California
  - Atlantis, Florida
  - Brooksville, Florida
  - Delray Beach, Florida
  - Fort Myers, Florida
  - Lake Worth, Florida
  - Miami, Florida
  - Orlando, Florida
  - St. Petersburg, Florida
  - Weston, Florida
  - Columbus, Georgia
  - Douglasville, Georgia
  - Chicago, Illinois
  - Park Ridge, Illinois
  - Baton Rouge, Louisiana
  - Bangor, Maine
  - Chestnut Hill, Massachusetts
  - Plymouth, Massachusetts
  - Flowood, Mississippi
  - Creve Coeur, Missouri
  - Princeton, New Jersey
  - Springfield, New Jersey
  - Brooklyn, New York
  - Latham, New York
  - New York, New York
  - Staten Island, New York
  - Wilmington, North Carolina
  - Columbus, Ohio
  - Portland, Oregon
  - Norristown, Pennsylvania
  - Philadelphia, Pennsylvania
  - San Antonio, Texas
  - Wichita Falls, Texas
  - Murray, Utah
  - Salt Lake City, Utah
  - Bennington, Vermont
  - Williamsburg, Virginia
- Australia (3):
  - Hornsby, New South Wales
  - Geelong, Victoria
  - West Heidelberg, Victoria
- Belgium (3):
  - Brussels
  - Leuven
  - Saint Truiden
- Canada (4):
  - Kelowna, British Columbia
  - Chatham, Ontario
  - Toronto, Ontario
  - Gatineau, Quebec
- France (4):
  - Nice
  - Paris
  - Rouen
  - Toulouse
- Germany (4):
  - Achim
  - Cologne
  - München
  - Nuremberg
- Italy (2):
  - Brescia, Brescia
  - Milan, Milano
- Mexico (2):
  - Guadalajara, Jalisco
  - Monterrey, Nuevo León
- Poland (4):
  - Bialystok
  - Bydgoszcz
  - Poznan
  - Warsaw
- South Africa (4):
  - Bellville
  - Johannesburg
  - Pretoria
  - Somerset West
- South Korea (3):
  - Seongnam-si, Gyenggi-go
  - Busan
  - Seoul
- Spain (5):
  - Elche, Altcante
  - Barcelona, Barcelona
  - Terrassa, Barcelona
  - Madrid, Madrid
  - Burgos